CLINICAL TRIAL: NCT00003825
Title: Phase III Study of Pentosanpolysulfate (PPS) in Treatment of GI Tract Sequelae of Radiotherapy
Brief Title: Pentosan Polysulfate in Treating Patients With Gastrointestinal Disturbance Caused by Radiation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: RTOG-9809; CDR0000066979
Record Dates: First submitted 1999-11-01; First posted 2004-05-03 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2013-08

CONDITIONS: Diarrhea; Radiation Enteritis
Keywords: radiation enteritis; diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Pentosan Sulfuric Polyester

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: pentosan polysulfate sodium
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Pentosan polysulfate may be effective in treating side effects of radiation therapy to the abdomen or pelvis. It is not yet known whether pentosan polysulfate is more effective than no further therapy for treating gastrointestinal disturbance caused by previous radiation therapy.

PURPOSE: Randomized phase III trial to determine the effectiveness of pentosan polysulfate in treating patients who have inflammation of the rectum, diarrhea, or blood in stools caused by previous radiation therapy to the abdomen and pelvis.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of pentosan polysulfate in patients with gastrointestinal tract sequelae after radiotherapy to the abdomen and pelvis. II. Determine the toxic effects of this drug in these patients. III. Determine the effect of this drug on symptoms and quality of life of these patients.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms. Arm I: Patients receive oral pentosan polysulfate three times a day for 2-6 months. Arm II: Patients receive oral placebo three times a day for 2-6 months. Both arms: Patients may receive retreatment for two months if symptoms return and last for at least 2 weeks. Quality of life is assessed before treatment, and at each follow up visit. Patients are followed every 2 months for 6 months, then every 3 months for 18 months, then annually for 3 years.

PROJECTED ACCRUAL: A total of 174 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Must have received prior radiotherapy to the abdomen and pelvis and now have radiation related gastrointestinal symptoms (which were not present before the radiotherapy and/or attributed to other causes) Proctitis Diarrhea Melena (blood in stools) Severity of symptoms classified as grade 1, 2, or 3

PATIENT CHARACTERISTICS: Age: Any age Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No bleeding ulcers No bleeding diathesis

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 1 month since prior chemotherapy No concurrent chemotherapy Endocrine therapy: Concurrent hormonal therapy for prostate cancer allowed Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy Surgery: No prior bowel resection At least 3 weeks since prior surgery Other: No concurrent anticoagulation therapy (except aspirin)

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 1999-06; Primary Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miljenko V. Pilepich, MD, Study Chair — Saint Joseph Mercy Cancer Center
Locations (260):
- United States (241):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Urology Associates - Mobile AL, Mobile, Alabama
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscaloosa, Alabama
  - Providence Cancer Therapy Center, Anchorage, Alaska
  - Arizona Cancer Center, Tucson, Arizona
  - Mount Diablo Medical Center, Concord, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - University of California San Diego Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Cancer Care Center, Pomona, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - Radiation Medical Group, Inc., San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Stanford University, Stanford, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Whittingham Cancer Center, Norwalk, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lykes Center for Radiation Therapy, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Radiation Therapy Associates - Fort Myers, Fort Myers, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Radiation Oncology Group, Orange Park, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - West Florida Cancer Institute - Pensacola, Pensacola, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - InterCommunity Cancer Center at Rome, Rome, Georgia
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Provena St. Joseph Hospital- Regional Cancer Care Center, Elgin, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Clarion Health Partners Inc., Indianapolis, Indiana
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - St. Joseph's Radiation Oncology Center, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Western Baptist Hospital, Paducah, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Romagosa Radiation Oncology Center, Lafayette, Louisiana
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Radiation Oncology Affiliates of Maryland, P.A., Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Saint Josephs Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Regional Medical Center, Midland, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's Medical Center, Saginaw, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - North Mississippi Medical Center/Cancer Center, Tupelo, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - Nebraska Health System, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Hospital - Millville, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua-Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Saint Joseph Medical Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Radiation Oncology, P.C., Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Catawba Memorial Hospital, Hickory, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Meritcare Roger Maris Cancer Center, Fargo, North Dakota
  - UNIMED Medical Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - St. John Medical Center, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Regional Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Catholic Medical Center, Mercy Fitzgerald Divison, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Penn State Geisinger Cancer Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Julie and Ben Rogers Cancer Institute, Beaumont, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - East Texas Medical Center - Cancer Institute, Tyler, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Green Mountain Oncology Group, Rutland, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - RMH Regional Canter Center, Harrisonburg, Virginia
  - Virginia Baptist Hospital, Lynchburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - St. Joseph's Hospital, Milwaukee, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - Southeastern Wisconsin Regional Cancer Center, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (19):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Universitaire de Sante de l'Estrie - Site Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Pilepich MV, Paulus R, St Clair W, Brasacchio RA, Rostock R, Miller RC. Phase III study of pentosanpolysulfate (PPS) in treatment of gastrointestinal tract sequelae of radiotherapy. Am J Clin Oncol. 2006 Apr;29(2):132-7. doi: 10.1097/01.coc.0000203758.77490.fd. PMID 16601430